CLINICAL TRIAL: NCT04098796
Title: Anti-PD-1 Antibody Combined With Chemotherapy as First-line Treatment of Serum AFP-elevated Gastric or Gastroesophageal Junction Adenocarcinoma: a Single-arm, Multicenter Phase II Study
Brief Title: PD-1 Antibody + XELOX in 1st Line Serum A-fetoprotein (AFP)-Elevated Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jingdong Zhang, Director, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-1-CT-Ⅱ-1st L-AFPGC
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma; AFP
Keywords: Gastric or gastroesophageal junction adenocarcinoma; AFP; PD-1; chemotherapy; first-line
MeSH Terms: interventions — spartalizumab; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Anti-PD-1 antibody＋XELOX (Experimental): Every patient will receive anti-PD-1 antibody (200 mg intravenous drip every 3 weeks) and XELOX regimen chemotherapy (Oxaliplatin 130 mg/m2, intravenous drip, d1; Capecitabine 1000mg/ kg, twice a day, orally, d1-14;every 21 days). Anti-PD-1 antibody will be administered until the disease progresses or lasts for two years. XELOX will be administered 6-8cycles，followed by capecitabine monotherapy, the course of treatment is determined by the investigators according to clinical practice.
  Interventions: Drug: Anti-PD-1 antibody; Drug: XELOX

INTERVENTIONS:
Drug: Anti-PD-1 antibody — Sintilimab will be administered 200 mg intravenous drip, every 3 weeks. Anti-PD-1 antibody will be administered until the disease progresses or lasts for two years.
Drug: XELOX — Oxaliplatin 130 mg/m2, intravenous drip, d 1; Capecitabine 1000mg/ kg, twice a day, orally, d1-14; Every 21 days. XELOX 6-8cycles，followed by capecitabine monotherapy, the course of treatment is determined by the investigators according to clinical practice.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of of anti-PD-1 antibody in combination with chemotherapy as first-line treatment in patients with unresectable, locally advanced recurrent or metastatic serum AFP-elevated gastric and gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
AFP-elevated gastric adenocarcinoma is a special type of gastric cancer, with the characteristics of high risk of liver and lymph node metastasis, poor therapeutic effect, and dismal prognosis.

This prospective study is a single-arm, multicenter phase II clinical study to evaluate the efficacy and safety of anti-PD-1 antibody in combination with chemotherapy as first-line treatment in patients with unresectable, locally advanced recurrent or metastatic serum AFP-elevated gastric and gastroesophageal junction adenocarcinoma.

AFP elevation is defined as serum AFP > 20 ng/ml. In this prospective study, the objective remission rate (ORR) will be used as primary outcome measures and 30 patients will be recruited. Anti-PD-1 antibody in combination with chemotherapy will be administered. PD-L1 expression and tumor mutant burden (TMB) will be measured before treatment. In addition, the dynamic changes of serum AFP levels, T lymphocyte in peripheral blood will be monitored during treatment. In the course of treatment, safety evaluation will be carried out according to the standard of adverse reaction classification (CTCAE) 4.0.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must volunteer to participate in the study, signed informed consent, and were able to comply with the program requirements of visits and related procedures.
2. Age and gender: ≥18 years old and≤75 years old, both men and women.
3. All subjects must have unresectable, local advanced recurrent or metastatic gastric adenocarcinoma (GC) or gastroesophageal junction adenocarcinoma (GEC) confirmed by histologically.
4. No systematic treatment for advanced or metastatic GC/GEC has been received in the past. For patients who have received adjuvant or neoadjuvant therapy (including chemotherapy, radiotherapy and/or radiochemotherapy) for GC/GEC in the past, the last treatment must be completed at least six months before the start of study drug. Subjects are allowed to receive palliative radiotherapy, but it must be completed two weeks before the start of study drug.
5. Serum AFP > 20 ng/ml.
6. All acute toxic reactions caused by previous medication or surgery were alleviated to grade 0-1 (according to NCI-CTCAE version 5.0) or to the level specified by the criteria for Inclusion/exclusion. The toxicities that do not pose a safety risk to patients determined by investigators are excluded, such as hair loss , etc.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
8. Expected survival: ≥12 weeks.
9. Subject must have at least one measurable lesion or evaluable disease by CT or MRI per RECIST 1.1 criteria.
10. The functions of important organs must meet the following requirements:(1)Hematological system: Neutrophil count≥1.5×10^9/L; Platelet count≥80×10^9/L; Hemoglobin≥90g/L;(2)Liver function: Serum albumin≥28g/L; Total bilirubin (TBI)≤1.5×ULN; Alanine aminotransferase (ALT)≤2.5×ULN (or≤5×ULN if liver metastases are present); Aspartate aminotransferase (AST)≤2.5×ULN (or≤5×ULN if liver metastases are present); (3)Renal function: Serum creatinine≤1.5×ULN or calculated creatinine clearance (CrCl) ≥40 mL/min (using the Cockcroft-Gault formula):Female CrCl = (140- age in years) × weight in kg × 0.85/ 72 × serum creatinine in mg/ dL; Male CrCl = (140- age in years) × weight in kg × 1.00/72 × serum creatinine in mg/ dL;(4)Coagulation function: Subjects not receiving anticoagulation therapy: (International Normalized Ratio) INR or activeated partial thromboplastin time (APTT) ≤ 1.5×ULN.
11. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days prior to the start of study drug. WOCBP must agree to follow instructions for method(s) of contraception (e.g. intrauterine devices, contraceptives, condoms or abstinence) for the duration of study treatment and 6 months after the last dose of study treatment. Subjects must be non-lactating. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment and 6 months after the last dose of study treatment.

Exclusion Criteria:

1. Known human epidermalgrowth factor receptor-2 (HER2) positive.
2. Currently participating in research and receiving research treatment, or participating in the research of experimental drugs within four weeks before the start of study drug, and having received research treatment or used experimental instruments.
3. Major surgery were performed within 4 weeks before the start of the study and incomplete recovery.
4. Existence of any active autoimmune disease or with a history of autoimmune disease (as the following examples, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary, vasculitis, nephritis, hyperthyroidism; patients with vitiligo; in childhood asthma has been completely alleviated, adults without any intervention can be included; asthma with medical intervention could not be included). Substitution therapy is not considered as systemic therapy. Patients with the following diseases are not excluded and may proceed to further screening: a. Controlled Type I diabetes; b. Hypothyroidism (provided it is managed with hormone replacement therapy only).
5. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 7 days before randomization.
6. Any active malignancy ≤ 5 years before randomization except for the specific cancer under investigation in this study and any cured limited tumors (eg, carcinoma in situ of the cervix or prostate, basal cell skin cancer).
7. Patients with known central nervous system metastasis (suspected need to be excluded by MRI scans) or a history of hepatic encephalopathy.
8. A history of pneumonia (non-infectious) requiring steroid therapy within 6 months or currently suffering from pneumonia (pulmonary infectious).
9. With active infections, fever of unknown origin (≥38.5℃) within 7 days before the start of study drug; or white blood cell count at baseline > 15×10^9/L); with severe chronic or active infections (including tuberculosis infection, etc.) requiring systemic antibacterial, antifungal or antiviral therapy during screening period, excluding viral hepatitis.
10. With any other disease, metabolic abnormality, abnormal physical examination or abnormal laboratory examination, according to the judgments of the investigators, there is reason to suspect that the patient has a certain disease or condition that is not suitable for the use of study drugs, or that it will affect the interpretation of research results or put the patient at high risk.
11. Mental or drug abuse disorders known to have an impact on compliance with study requirements
12. Congenital or acquired immunodeficiency (e.g. HIV-infected persons).
13. With active hepatitis B virus (HBV) or hepatitis C virus (HCV). Active hepatitis B is defined as known positive HBsAg results, and HBV-DNA > 2000IU/ml. Active hepatitis C is defined as known positive hepatitis C antibodies and the quantitative results of HCV RNA are higher than the lower detection limit of analytical methods. Active HBV will be allowed if they have HBV DNA < 500 IU/mL (or 2500 copies/mL) at screening. Patients with HBV-DNA < 2000IU/ml through antiviral therapy can be considered included.
14. Was administered a live attenuated vaccine ≤ 4 weeks before randomization, or plan to vaccinate during treatment with against PD-1 monoclonal antibody or within five months after last administration.
15. More than a small amount of pericardial effusion, uncontrolled pleural effusion or clinically obvious peritoneal effusion at screening. It is defined as meeting the following criteria: physical examination at screening can detect pleural and peritoneal effusion, or in screening process, pleural and peritoneal effusion needs puncture and drainage.
16. With history of serious cardiovascular and cerebrovascular diseases: (1) Any history of heart failure meeting New York Heart Association Classification III or IV or more serious history of heart disease, myocardial infarction, or cerebrovascular accident in 3 months before randomization；(2) Left ventricular ejection fraction < 50% by color Doppler echocardiography；(3) Uncontrollable hypertension; (4) Uncontrolled arrhythmias; (5) Acute coronary syndrome, congestive heart failure, stroke, thromboembolism or other cardiovascular events above grade 3 within 6 months before the start of study drug.
17. A history of allergy to anti-PD-1, anti-PD-L1 monoclonal antibody drugs or oxaliplatin or capecitabine.
18. Known dihydropyrimidine dehydrogenase deficiency.
19. Pregnant or lactating women; or female subjects who are expected to conceive during the planned trial period (from the start of screening visits to 120 days after the last administration of the study) or male subjects whose spouses are pregnant.
20. Other situations that the researchers think should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The proportion of patients whose best overall response (BOR) is complete response (CR) or partial response (PR) assessed by RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  The time from the date of randomization to the date of first documentation of disease progression or death, whichever occurs first.
Overall survival (OS) | 2 years
  The time from the date of randomization until the date of death due to any cause.
Duration of response (DOR) | 2 years
  The time from CR or PR to disease progression or death.
Disease control rate (DCR) | 2 years
  The proportion of patients who's BOR is CR, PR, and stable disease (SD) assessed.
6-month/9-month/12-month survival rate | 6-month/9-month/12-month
  After date of randomization, evaluate patient survival rate at 6,9 and 12 months, respectively.
Incidence of Treatment-Emergent Adverse Events | 2 years
  Incidence of Treatment-Emergent Adverse Events.The grade of toxicity will be assessed using the NCI-CTCAE version 5.0.
Quality of life score (QLQ-C30) | Every 2 weeks after the first treatment until 2 years
  Scores according to the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 scoring manual.
Exploration of biomarkers (PD-L1 expression, TMB at the baseline, changes of AFP and T lymphocyte in peripheral blood) | 2 years
  PD-L1 expression at the baseline using, TMB level at the baseline, changes of serum AFP level and T lymphocyte in peripheral blood at baseline and during the treatment，and etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jingdong Zhang, Principal Investigator — China Medical University, China
Locations (1):
- Liaoning Cancer Hospital & Institute, Shenyang, Liaoning, China